CLINICAL TRIAL: NCT03068676
Title: A Pilot Study Investigating the Feasibility of Implementing Internet-delivered Treatments for Depression and Anxiety in Primary Care
Brief Title: Internet-delivered Treatments for Depression and Anxiety in Primary Care (SUMMA)
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Paused due to technical issues
Sponsor: Silver Cloud Health (Other)
Collaborators: Summa Health System (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SUMMA-PC
Record Dates: First submitted 2017-02-21; First posted 2017-03-03 (Actual); Last update posted 2018-09-10 (Actual); Status verified 2018-09

CONDITIONS: Depressive Disorder; Anxiety Disorders; Depression
Keywords: Depression; Anxiety; Internet-delivered; CBT; Primary Care
MeSH Terms: conditions — Depressive Disorder; Anxiety Disorders; Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Space from depression (Experimental): Space from Depression is an eight-module online CBT-based intervention for depression, composed of cognitive and behavioral components including self-monitoring and thought recording, behavioral activation, cognitive restructuring, and challenging core beliefs. Each module follows a structured format that incorporates introductory quizzes, videos, informational content, interactive activities, as well as homework suggestions and summaries. In addition, personal stories and accounts from other users are incorporated into the presentation of the material.
  Interventions: Behavioral: Space from Depression
- Space from Anxiety (Experimental): Space from Anxiety is an eight-module online CBT-based intervention for depression, composed of cognitive and behavioral components including self-monitoring and thought recording, behavioral activation, cognitive restructuring, and challenging core beliefs. Each module follows a structured format that incorporates introductory quizzes, videos, informational content, interactive activities, as well as homework suggestions and summaries. In addition, personal stories and accounts from other users are incorporated into the presentation of the material.
  Interventions: Behavioral: Space from Anxiety

INTERVENTIONS:
Behavioral: Space from Depression — internet-delivered CBT
  Arms: Space from depression
Behavioral: Space from Anxiety — internet-delivered CBT
  Arms: Space from Anxiety

SUMMARY:
The current study is an open feasibility trial with the aim of providing a description of the factors associated with the implementation of an iCBT platform into an existing treatment framework in a primary care setting. The trial will examine the factors surrounding implementation, such as the experience of primary care practitioners and the online supporters, the recruitment process, and attitudes towards the overall implementation of the interventions. Patients presenting to the primary care setting will be screened using standard depression and anxiety measures, and where appropriate, will be referred to an iCBT intervention for either depression or anxiety, with support from trained staff. Analyses will be conducted on outcome measures to examine changes in symptom severity as patients progress through the intervention. Patient satisfaction data will also be collected to establish patient acceptability of the intervention. [Note: Recruitment is ONLY open to patients at Ohio Family Practice Center]

DETAILED DESCRIPTION:
iCBT is the delivery of a tailored structured cognitive and behaviour therapy based programme, with support, to individuals with mild to moderate symptoms of depression and anxiety. There is now a substantial body of research evidence that supports the efficacy and effectiveness of internet-delivered cognitive behaviour therapy for depression and anxiety. Historically, a number of iCBT interventions have been used in clinical practice in IAPT services. However, they have often suffered with poor engagement and consequently poor clinical outcomes. More recent developments in the field have produced more robust technological platforms, where content is delivered through a variety of media that enhance productivity, increase engagement and produce better clinical outcomes. The SilverCloud intervention has been demonstrated to be a clinical effective evidence-based cognitive behavioural treatment option.

Approximately 90% of primary care patients with depression have one or more visits to a primary care physician (PCP) over a 12-month period, whereas less than one-third see a mental health professional. It has been reported that individuals with an anxiety disorder are 3 to 5 times more likely to visit their primary care physician than those without, but their symptoms are often associated with physical causes. PCPs often do not have training in psychological therapies and therefore they do not feel competent to treat individuals presenting with depression or anxiety. Often these individuals are prescribed antidepressant or anti-anxiety medications.

The use of online programs to deliver CBT to people with mental health disorders is becoming increasingly popular. Internet-delivered CBT (iCBT) consists of programs designed for the treatment of specific disorders, such as depression and anxiety, which are delivered via the internet. These programs can be clinician-guided and/or self-administered interventions. Evidence suggests that iCBT can benefit individuals with anxiety and depression when offered in a service context that offers brief support from trained staff. Such iCBT interventions are widely-used in some European countries and the recommended length of treatment is generally 6 - 8 online sessions. A robust evidence base supporting the use and effectiveness of internet-delivered treatments for depression and anxiety has been established. Outcomes have been greater for those programs offering the additional feature of human support.

The current study will examine the feasibility of implementing an iCBT platform within a primary care setting. This objective can be further dismantled into several sub objectives:

1. Is the model of implementation (screening, recruitment, and adherence to the internet-delivered intervention) feasible?
2. Will patients experience the iCBT intervention as satisfactory within their primary care treatment?
3. What is the feedback of the Primary Care Practitioners about the implementation of the internet-delivered intervention as part of primary care?
4. What is the experience of the trained supporters who assist patients within the iCBT intervention?
5. Can an internet-delivered intervention achieve improvements in depressive and anxiety symptoms for users?
6. Can patient attitudes toward internet-delivered interventions predict treatment outcome?

ELIGIBILITY:
Inclusion criteria:

At least 18 years of age, Speak English, Self-report symptoms of depression or anxiety (using PHQ-9 and GAD-7 measures).

Specifically for the self-report symptoms,

participants will need to have a PHQ-9 score of 5 to 19 for the depression program or a GAD-7 score of 5 to 15 for the anxiety program.

Participants currently attending face-to-face therapy/counseling will be excluded.

Exclusion criteria

Participants who flag as a risk on the self-harm item of the PHQ-9 during routine office visit screening will not be referred to the study and will be provided treatment and/or referral services as per the clinic's standard procedure.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2017-02-08 (Actual); Primary Completion 2018-02-08 (Actual); Study Completion 2018-02-09 (Actual)

PRIMARY OUTCOMES:
Patient health Questionnaire | At week 8
  The PHQ-9 is a self-report measure of depression that has been widely used in screening, primary care, and research. The PHQ-9 items reflect the diagnostic criteria for depression outlined by the Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition - Text Revision (DSM-IV-TR) (American Psychiatric Association [APA], 2000). Summed scores range from 0-27; larger scores reflect a greater severity of depressive symptoms. The PHQ-9 discriminated well between depressed and nondepressed individuals using the clinical cut-off of total score ≥10, with good sensitivity (88.0%) and specificity (88.0%) (Kroenke et al., 2001; R. Spitzer et al., 1999).
Generalized Anxiety Disorder | At week 8
  The GAD-7 (Spitzer, Krownke, Williams, & Lowe, 2006) comprises 7 items measuring symptoms and severity of GAD based on the DSM-IV diagnostic criteria for GAD. The GAD-7 has good internal consistency (.89) and good convergent validity with other anxiety scales. Higher scores indicate greater severity of symptoms. The GAD-7 is increasingly used in large-scale studies as a generic measure of changes in anxiety symptomatology, using a cut-off score of 8 (Richards & Suckling, 2009).

SECONDARY OUTCOMES:
Socio-demographic Questionnaire | At baseline for screening
  Collects information on the characteristics of the sample including age, gender etc.
Work and Social Adjustment | At baseline and week 8
  The Work and Social Adjustment (WASA; Mundt, Marks, Shear, & Greist, 2002) is a simple, reliable and valid measure of impaired functioning. It is a simple and reliable (α >.75) 5-item self-report measure that provides an experiential impact of a disorder from the patient's point of view. It looks at how the disorder impairs the patient's ability to function day to day on five dimensions: work, social life, home life, private life and close relationships.
Satisfaction with Treatment | At week 8
  The Satisfaction with Treatment (SAT; Timulak & Richards, 2012) measure contains several questions that aim to assess patient satisfaction with the iCBT intervention received. The measure consists of 2 qualitative questions and several quantitative questions, centring on what the patients liked or disliked about the iCBT intervention.
Attitudes towards Psychological Online Interventions | At baseline and week 8
  The Attitudes towards Psychological Online Interventions (APOI; Schroder et al., 2015) will be administered to patients at both pre and post intervention time points. The APOI is a brief inventory that assesses attitudes towards online interventions across four domains - scepticism and perception of risks, confidence in effectiveness, technologization threat and anonymity benefits.

CONTACTS AND LOCATIONS:
Overall Officials: Derek Richards, PhD, Study Director — SilverCloud Health
Locations (1):
- Summa Health, Akron, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Andersson G, Cuijpers P. Internet-based and other computerized psychological treatments for adult depression: a meta-analysis. Cogn Behav Ther. 2009;38(4):196-205. doi: 10.1080/16506070903318960. PMID 20183695
- [Background] Coyne JC, Fechner-Bates S, Schwenk TL. Prevalence, nature, and comorbidity of depressive disorders in primary care. Gen Hosp Psychiatry. 1994 Jul;16(4):267-76. doi: 10.1016/0163-8343(94)90006-x. PMID 7926703
- [Background] Faul F, Erdfelder E, Lang AG, Buchner A. G*Power 3: a flexible statistical power analysis program for the social, behavioral, and biomedical sciences. Behav Res Methods. 2007 May;39(2):175-91. doi: 10.3758/bf03193146. PMID 17695343
- [Background] Goldman LS, Nielsen NH, Champion HC. Awareness, diagnosis, and treatment of depression. J Gen Intern Med. 1999 Sep;14(9):569-80. doi: 10.1046/j.1525-1497.1999.03478.x. PMID 10491249
- [Background] Hedman E, Ljotsson B, Lindefors N. Cognitive behavior therapy via the Internet: a systematic review of applications, clinical efficacy and cost-effectiveness. Expert Rev Pharmacoecon Outcomes Res. 2012 Dec;12(6):745-64. doi: 10.1586/erp.12.67. PMID 23252357
- [Background] Katon WJ, Roy-Byrne P, Russo J, Cowley D. Cost-effectiveness and cost offset of a collaborative care intervention for primary care patients with panic disorder. Arch Gen Psychiatry. 2002 Dec;59(12):1098-104. doi: 10.1001/archpsyc.59.12.1098. PMID 12470125
- [Background] Kessler RC, McGonagle KA, Zhao S, Nelson CB, Hughes M, Eshleman S, Wittchen HU, Kendler KS. Lifetime and 12-month prevalence of DSM-III-R psychiatric disorders in the United States. Results from the National Comorbidity Survey. Arch Gen Psychiatry. 1994 Jan;51(1):8-19. doi: 10.1001/archpsyc.1994.03950010008002. PMID 8279933
- [Background] Khouzam, H. R. (2009). Anxiety Disorders: Guidelines for Effective Primary Care, Part 1, Diagnosis. Consultant, 49 (3).
- [Background] Kohn R, Saxena S, Levav I, Saraceno B. The treatment gap in mental health care. Bull World Health Organ. 2004 Nov;82(11):858-66. Epub 2004 Dec 14. PMID 15640922
- [Background] Kroenke K, Spitzer RL, Williams JB. The PHQ-9: validity of a brief depression severity measure. J Gen Intern Med. 2001 Sep;16(9):606-13. doi: 10.1046/j.1525-1497.2001.016009606.x. PMID 11556941
- [Background] Kroenke K, Spitzer RL, Williams JB, Monahan PO, Lowe B. Anxiety disorders in primary care: prevalence, impairment, comorbidity, and detection. Ann Intern Med. 2007 Mar 6;146(5):317-25. doi: 10.7326/0003-4819-146-5-200703060-00004. PMID 17339617
- [Background] Lecrubier Y, Weiller E. Characteristics, recognition and treatment of dysthymics in primary care. Eur Psychiatry. 1998 Jul;13(4):198-202. doi: 10.1016/S0924-9338(98)80004-7. PMID 19698625
- [Background] Lepine JP. The epidemiology of anxiety disorders: prevalence and societal costs. J Clin Psychiatry. 2002;63 Suppl 14:4-8. PMID 12562112
- [Background] Lyness JM, Caine ED, King DA, Cox C, Yoediono Z. Psychiatric disorders in older primary care patients. J Gen Intern Med. 1999 Apr;14(4):249-54. doi: 10.1046/j.1525-1497.1999.00326.x. PMID 10203638
- [Background] Mohr DC, Ho J, Duffecy J, Baron KG, Lehman KA, Jin L, Reifler D. Perceived barriers to psychological treatments and their relationship to depression. J Clin Psychol. 2010 Apr;66(4):394-409. doi: 10.1002/jclp.20659. PMID 20127795
- [Background] Musiat P, Goldstone P, Tarrier N. Understanding the acceptability of e-mental health--attitudes and expectations towards computerised self-help treatments for mental health problems. BMC Psychiatry. 2014 Apr 11;14:109. doi: 10.1186/1471-244X-14-109. PMID 24725765
- [Background] Richards D, Richardson T. Computer-based psychological treatments for depression: a systematic review and meta-analysis. Clin Psychol Rev. 2012 Jun;32(4):329-42. doi: 10.1016/j.cpr.2012.02.004. Epub 2012 Feb 28. PMID 22466510
- [Background] Richards D, Timulak L, O'Brien E, Hayes C, Vigano N, Sharry J, Doherty G. A randomized controlled trial of an internet-delivered treatment: Its potential as a low-intensity community intervention for adults with symptoms of depression. Behav Res Ther. 2015 Dec;75:20-31. doi: 10.1016/j.brat.2015.10.005. Epub 2015 Oct 21. PMID 26523885
- [Background] Richards DA, Suckling R. Improving access to psychological therapies: phase IV prospective cohort study. Br J Clin Psychol. 2009 Nov;48(Pt 4):377-96. doi: 10.1348/014466509X405178. Epub 2009 Feb 9. PMID 19208291
- [Background] Schulberg HC, Mulsant B, Schulz R, Rollman BL, Houck PR, Reynolds CF 3rd. Characteristics and course of major depression in older primary care patients. Int J Psychiatry Med. 1998;28(4):421-36. doi: 10.2190/G23R-NGGN-K1P1-MQ8N. PMID 10207741
- [Background] Sheehan DV. Depression: underdiagnosed, undertreated, underappreciated. Manag Care. 2004 Jun;13(6 Suppl Depression):6-8. PMID 15293765
- [Background] Simon GE, Goldberg D, Tiemens BG, Ustun TB. Outcomes of recognized and unrecognized depression in an international primary care study. Gen Hosp Psychiatry. 1999 Mar-Apr;21(2):97-105. doi: 10.1016/s0163-8343(98)00072-3. PMID 10228889
- [Background] Spek V, Cuijpers P, Nyklicek I, Riper H, Keyzer J, Pop V. Internet-based cognitive behaviour therapy for symptoms of depression and anxiety: a meta-analysis. Psychol Med. 2007 Mar;37(3):319-28. doi: 10.1017/S0033291706008944. Epub 2006 Nov 20. PMID 17112400
- [Background] Spitzer RL, Kroenke K, Williams JB. Validation and utility of a self-report version of PRIME-MD: the PHQ primary care study. Primary Care Evaluation of Mental Disorders. Patient Health Questionnaire. JAMA. 1999 Nov 10;282(18):1737-44. doi: 10.1001/jama.282.18.1737. PMID 10568646
- [Background] Spitzer RL, Kroenke K, Williams JB, Lowe B. A brief measure for assessing generalized anxiety disorder: the GAD-7. Arch Intern Med. 2006 May 22;166(10):1092-7. doi: 10.1001/archinte.166.10.1092. PMID 16717171
- [Background] Spitzer RL, Williams JB, Kroenke K, Linzer M, deGruy FV 3rd, Hahn SR, Brody D, Johnson JG. Utility of a new procedure for diagnosing mental disorders in primary care. The PRIME-MD 1000 study. JAMA. 1994 Dec 14;272(22):1749-56. PMID 7966923
- [Background] Stein MB, McQuaid JR, Pedrelli P, Lenox R, McCahill ME. Posttraumatic stress disorder in the primary care medical setting. Gen Hosp Psychiatry. 2000 Jul-Aug;22(4):261-9. doi: 10.1016/s0163-8343(00)00080-3. PMID 10936633
- [Background] Vermani M, Marcus M, Katzman MA. Rates of detection of mood and anxiety disorders in primary care: a descriptive, cross-sectional study. Prim Care Companion CNS Disord. 2011;13(2):PCC.10m01013. doi: 10.4088/PCC.10m01013. PMID 21977354
- [Background] Wang PS, Lane M, Olfson M, Pincus HA, Wells KB, Kessler RC. Twelve-month use of mental health services in the United States: results from the National Comorbidity Survey Replication. Arch Gen Psychiatry. 2005 Jun;62(6):629-40. doi: 10.1001/archpsyc.62.6.629. PMID 15939840
- [Background] Williams JW Jr, Mulrow CD, Kroenke K, Dhanda R, Badgett RG, Omori D, Lee S. Case-finding for depression in primary care: a randomized trial. Am J Med. 1999 Jan;106(1):36-43. doi: 10.1016/s0002-9343(98)00371-4. PMID 10320115